CLINICAL TRIAL: NCT01256749
Title: A Comparative Study of Global 12 Lead Electroencephalogram to Frontal SedlineTM Electroencephalogram Monitoring for the Evaluation of Intraoperative Burst Suppression During Elective Craniotomy or Transphenoidal Pituitary Resection
Brief Title: A Comparative Study of Global 12 Lead Electroencephalogram to Frontal SedlineTM Electroencephalogram
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Deborah McIvor, MD, MD, Loma Linda University
Other Study IDs: 5100294
Record Dates: First submitted 2010-12-02; First posted 2010-12-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Craniotomy; Transphenoidal Pituitary Resection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The fundamental reason for comparing the ability of the Frontal Sedline TM Electroencephalogram (PSA EEG) to standard Global 12 Lead Electroencephalogram (EEG) for burst suppression detection is to determine if a less expensive, less invasive and possibly more convenient bifrontal EEG monitor can be effective for evaluation of anesthesia-induced intraoperative burst suppression therapy (IBST) for cerebral protection.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ASA class 1-3 male or female 18-90 years of age;
2. scheduled for elective craniotomy in the LLUMC University Hospital, for which the surgeon has requested intraoperative burst suppression therapy;
3. capable of understanding and signing informed consent;
4. willing to have dual EEG monitoring.

Exclusion Criteria:

1. Age under 18 years;
2. emergency or trauma situation requiring craniotomy;
3. surgical approach that prohibits placing the SEDLineTM array on the forehead;
4. known sensitivity to the adhesives on the SEDLineTM array;
5. lack of availability of standard EEG monitoring;
6. patients with seizure disorders and refusal of consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective craniotomy or transphenoidal pituitary resection at LLUMC University Hospital in which the surgeon has requested intraoperative burst suppression therapy regardless of the inciting etiology will be eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Correlation between 4 channel PSA EEG and a global 12 lead EEG | 24 hours
  The primary outcome measure is correlation between 4 channel frontal PSA EEG pattern and standard global 12 lead EEG during IBST.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah W McIvor, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States